CLINICAL TRIAL: NCT02179099
Title: Pilot Study Evaluating Safety and Efficacy of Intravesical Instillations of Botulinum Toxin in TC-3 Gel in OAB Patients
Brief Title: Safety and Efficacy of Intravesical Botulinum Toxin in TC-3 Gel in OAB Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Decision to open a randomized controlled trial with two groups receiving different Botulinum Toxin in comparison to placebo group.
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TC-OAB-02
Record Dates: First submitted 2014-06-29; First posted 2014-07-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; OAB; urgency; botulinum toxin; BTX; botox; intravesical; TheraCoat; TCGel; TC-3 Gel
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BTX mixed with TC-3 Gel (Experimental): Patients will be treated with a single intravesical instillation of 40 ml TC-3 gel mixed with 300U BTX
  Interventions: Device: BTX mixed with TC-3 Gel

INTERVENTIONS:
Device: BTX mixed with TC-3 Gel — Patients will be treated with a single intravesical instillation of 40 ml TC-3 gel mixed with 300U BTX
  Other Names: TCGel; TheraCoat hydrogel; Botox; botulinum toxin A; BTX

SUMMARY:
This is a single arm pilot study evaluating the feasibility and preliminary safety of a single intravesical instillation of TC-3 gel mixed with botulinum toxin (BTX) for symptomatic improvement in overactive bladder patients.

DETAILED DESCRIPTION:
BTX is considered as therapeutic option for overactive bladder (OAB). Randomized placebo-controlled studies have shown that BTX administered by intramural injection into the bladder wall in patients with OAB leads to significant improvement in urodynamic parameters and quality of life. (Schurch 2008). On the other hand, the animal study suggests that intravesically applied BTX acts to decrease frequency of bladder contraction by inhibiting sensory mechanism in the urothelium rather than directly through inhibition of the smooth muscle contraction. (Khera 2005). The efficacy of intravesical BTX instillation was only tested in a few open label trials for overactive bladder patients whereby the clinical improvement observed was short-lasting with a mean duration of 6.8 weeks (Petrou 2009, Krhut 2011). The short exposure duration of the urothelium to BTX could be one of the factors responsible for the lack of a sustained effect. TC-3 is a hydrogel with reverse thermal gelation properties that when mixed with BTX and instilled intravesically serves as the drug reservoir allowing for gradual release of BTX and thereby for its extended contact with bladder urothelium.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 to 85 years old with symptoms of idiopathic OAB for ≥ 3 months prior to screening.
* Patient has signed Informed Consent Form and is willing and able to comply with all requirements of the protocol, including proper completion of the voiding diaries and self-administered questionnaires.
* Patient is non-responder to anticholinergic or beta-agonist drug therapy or is not compliant to the treatment due has intolerable side effects.
* Patient has urination frequency of at least 8 micturitions per 24 hours.
* Patients has at least 3 urinary urgency incontinence (UUI) episodes per 3-day bladder diary, with no more than 1 incontinence-free day.
* Patients has PVR ≤100 ml. Patient with a single PVR of >100 ml and followed by two consecutive PVR measurements of <100 ml may be included in the study).
* If patient is a female of childbearing potential, she has a negative urine pregnancy test at screening visit and practice a reliable method of contraception throughout the study, until 6 months post treatment.
* Patient is mentally competent with the ability to understand and comply with the requirements of the study.
* Patient does not have active urinary tract infection as confirmed by urine culture. In case of UTI proven by urine culture, the patient will be treated with full course of antibiotics, and the instillation will be postponed for 1 week following negative urine culture demonstration.

Exclusion Criteria:

* Pregnant (positive urine pregnancy test), planning to become pregnant during the study period, breast-feeding, or of childbearing potential and not practicing reliable contraception**.
* Patient has a clinically significant Bladder Outlet Obstruction (BOO).
* Patient has neurogenic bladder.
* Patient currently uses Clean Intermittent Catheterization (CIC).
* Patient has documented unstable diabetes with or without diabetic neuropathy.
* Patient who is currently undergoing biofeedback, pelvic muscle rehabilitation, pelvic floor physical therapy, or electrical-stimulation.
* Patient with 24-hour total urine volume voided greater than 3,000 ml as measured at screening period.
* Patient with vesico-ureteral reflux, interstitial cystitis, genitourinary fistulae
* Patient with pelvic organ prolapse stage III or IV, (i.e. the most distal part of the prolapse protruding more than 1 cm beyond the hymen at straining)
* Patient with lower tract genitourinary malignancies
* Patient with prior anti-incontinence surgery and interventions including mid-urethral slings, Burch bladder suspension, sacral neuromodulation, or tibial nerve stimulation.
* Patient with prior Botox anti-incontinence therapy.
* Patient with previous pelvic radiation therapy
* Patient who is morbidly obese (BMI > 40 Kg/m2).
* Patient had been treated for 2 or more UTIs within last 6 months.
* Patient on immunomodulatory therapy (suppressive or stimulatory)
* Patient participated in prior clinical trials with BTX+TC-3 gel
* Patient has current major psychiatric disorder or other psychiatric or medical issues that would interfere with study participation (e.g. dementia, psychosis, upcoming major surgery, etc).
* Subject has severe cardiac, pulmonary, renal, or hepatic disease that in the judgment of the study physician would preclude participation in this study.
* Patient with a life expectancy of less than 12 months.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety | 16 weeks
  1. Adverse events measured during entire study period. Adverse events will be graded according to the Common Toxicity Criteria on a scale of 0 to 5.
  2. Presence of the urinary retention defined as a PVR >200 ml.
Efficacy | 16 weeks
  1. Number of urinary urge episodes in 24-hour period per 3-day voiding diary (primary endpoint - week 12 post instillation)
  2. Proportion of patients who had positive treatment response per Treatment Benefit Scale (TBS) (primary endpoint - week 12 post instillation).

SECONDARY OUTCOMES:
exploratory efficacy | 16 weeks
  1. Number of voids in 24-hour period per 3-day voiding diary (primary endpoint - week 12 post instillation)
  2. Number of urge incontinence episodes in 24-hour period per 3-day voiding diary (primary endpoint - week 12 post instillation)
  3. Number of nocturnal voids per night per 3-day voiding diary (primary endpoint - week 12 post instillation).
  4. Post Void Residual Volume (PVR) as measured by bladder ultrasonography (primary endpoint - week 12 post instillation)
  5. KHQ score (Kings Health Questionnaire) (primary endpoint - week 12 post instillation).
  6. I-QOL score (Incontinence Quality of Life questionnaire) (primary endpoint - week 12 post instillation).

CONTACTS AND LOCATIONS:
Overall Officials: Ami Sidi, Prof MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- Urology Department, Edith Wolfson Medical Center, Holon, Israel